CLINICAL TRIAL: NCT01606514
Title: Web-based Intervention for Disaster-Affected Youth and Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01MH081056-01A1 (NIH); 1R01MH081056-01A1 (NIH)
Record Dates: First submitted 2012-05-21; First posted 2012-05-25 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2012-08

CONDITIONS: Mental Health Wellness 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Child, Parenting, & Parent Web-Intervention (Experimental): Bounce Back Now Child, Parenting, & Parent Psychoeducation & Self-Help Web-Intervention.
  Interventions: Behavioral: Bounce Back Now Website
- Child & Parenting Web-Intervention (Experimental): Bounce Back Now Child & Parenting Psychoeducation and Self-Help Web-Intervention.
  Interventions: Behavioral: Bounce Back Now Website
- Child & Parent Web-based Assessment (No Intervention): Bounce Back Now Web-Based Symptom Assessment

INTERVENTIONS:
Behavioral: Bounce Back Now Website — Bounce Back Now is a web-based psychoeducation and self-help website
  Arms: Child & Parenting Web-Intervention; Child, Parenting, & Parent Web-Intervention

SUMMARY:
A single disaster, terrorist attack, or other large-scale incident can adversely affect thousands of youth and families. Immediate consequences may include unmet basic needs and high economic burden, particularly among underserved populations. Disasters also can dramatically affect family roles and relationships over time (e.g., family routines, marital stress, parent-child interactions). Whereas most youth are resilient in the aftermath of disasters (i.e., do not develop serious mental health or health-risk problems), the prevalence of various problems of public health significance (e.g., PTSD, depression, substance abuse) clearly increases in this population. This underscores the need for effective, widely accessible, culturally-appropriate and cost-efficient interventions that foster resilience or rapid recovery relative to the health effects of disasters. Yet, few evidence-informed resources are available to youth and families to facilitate post-disaster resilience and recovery. Primary aims of this project are: (a) to develop a Web-based intervention for disaster-affected adolescents and parents targeting prevalent health-related correlates of disasters (i.e., development phase), (b) to conduct a randomized controlled population-based study to examine feasibility and preliminary efficacy of the intervention (i.e., randomized controlled trial [RCT] phase) and cultural relevance (i.e., perceived applicability of the intervention to one's cultural group), and (c) to refine the intervention based on RCT-phase data.

ELIGIBILITY:
Inclusion Criteria:

* adolescent between the ages of 12-17 and primary caregiver,
* residence in study identified location(s) at time of disaster,
* home internet connectivity

Exclusion Criteria:

* adolescent's primary caregiver not available,
* no adolescents in home,
* not residing in location at time of disaster,
* poor or no internet connectivity

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2010-12; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in adolescent mental health symptoms | baseline, 4 month followup, and 12 month followup
Change in parent mental health symptoms | baseline, 4 month followup, 12 month followup
Change in parent-child conflict | baseline, 4 month followup, 12 month followup
Change in parent-child relationship quality | baseline, 4 month followup, 12 month followup

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Ruggiero, PhD, Principal Investigator — Medical University of South Carolina

REFERENCES:
- [Derived] Ruggiero KJ, Price M, Adams Z, Stauffacher K, McCauley J, Danielson CK, Knapp R, Hanson RF, Davidson TM, Amstadter AB, Carpenter MJ, Saunders BE, Kilpatrick DG, Resnick HS. Web Intervention for Adolescents Affected by Disaster: Population-Based Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2015 Sep;54(9):709-17. doi: 10.1016/j.jaac.2015.07.001. Epub 2015 Jul 11. PMID 26299292